CLINICAL TRIAL: NCT01990404
Title: Efficacy of Premixed Nitrous Oxide and Oxygen in Elderly Patient With Out-of-hospital Severe Acute Pain: a Randomized Double-blind Study
Brief Title: Efficacy of Premixed Nitrous Oxide and Oxygen in Elderly Patient With Out-of-hospital Severe Acute Pain
Acronym: MEOPA-PA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: inadequate recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/12/066; 2012-004129-25 (EudraCT Number)
Record Dates: First submitted 2013-09-27; First posted 2013-11-21 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Pain Acute
Keywords: Premixed nitrous oxide and oxygen; Severe acute pain; Prehospital setting
MeSH Terms: conditions — Acute Pain | interventions — Nitrous Oxide; Oxygen; Meopa; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premixed 50% nitrous oxide and oxygen (Active Comparator): The patient will be taken care by the physician SMUR or home emergency. Upon acceptance of participation in the study, the clock will be started at the time of the establishment of the face mask. Premixed 50% nitrous oxide and oxygen is administered for 30 minutes and an opioid titration is started 10 minutes after the introduction of gas, unless the patient expresses pain score EN <3/10.
  Interventions: Drug: Premixed 50% nitrous oxide and oxygen
- Medical air (Placebo Comparator): The patient will be taken care by the physician SMUR or home emergency. Upon acceptance of participation in the study, the clock will be started at the time of the establishment of the face mask. The medical air is administered for 30 minutes and an opioid titration is started 10 minutes after the introduction of gas, unless the patient expresses pain score EN <3/10.
  Interventions: Drug: Medical Air

INTERVENTIONS:
Drug: Premixed 50% nitrous oxide and oxygen — Premixed 50% nitrous oxide and oxygen is a gas in cylinder of 5 litres delivered by a face mask. The gases of the study are contained in anonymous bottles of the same capacity. Bottles will only be differentiated by a letter: A or B.
  Other Names: MEOPA
  Arms: Premixed 50% nitrous oxide and oxygen
Drug: Medical Air — Medical air is a gas in cylinder of 5 litres delivered by a face mask. The gases of the study are contained in anonymous bottles of the same capacity. Bottles will only be differentiated by a letter: A or B
  Arms: Medical air

SUMMARY:
Pain in the elderly is poorly evaluated and clearly under treated. Premixed nitrous oxide and oxygen is used in the emergency medical care of the trauma, burns, during transport of patient with pain. None randomized study has validated the use of premixed nitrous oxide and oxygen in the emergency department in the elderly. The aim of the study is to demonstrate the efficacy of premixed nitrous oxide and oxygen compared to medical air in elderly patient with out-of-hospital severe acute pain

DETAILED DESCRIPTION:
The primary endpoint is the percentage of patients with pain relief (with a numerical rating scale of 3/10 or lower) 15 minutes after randomisation. Secondary endpoints are treatment safety and adverse events, time to analgesia and duration of analgesia. This study will expect 108 patients assigned in two parallel groups, defined by a randomization scheme. Four sites will participate to the research. Eligible patients with a numeric rating scale (NRS) score higher than 6/10 are randomly allocated to receive either MEOPA, or medical air. Neither the investigator nor the nurse knows the treatment. Pain score will be measured at baseline and every 5 minutes until pain relief will be obtained. The safety evaluation will include non invasive monitoring of blood pressure, heart rate, and oxygen saturation by pulse oximetry (SpO2) and adverse events collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years old and over
* Severe acute pain (NRS score greater than 6)

Exclusion Criteria:

* Contraindication of premixed 50% nitrous oxide and oxygen

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percentage of patients with pain relief (with a numerical rating scale of 3/10 or lower) | 15 minutes after randomisation

SECONDARY OUTCOMES:
adverse events | From the randomization until 48 hours after randomization
time to analgesia | From randomization until 48 hours
Duration of analgesia. | From randomization until 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bounes, MD, Principal Investigator — University Hospital of Toulouse
Locations (3):
- France (2):
  - SAMU Bobigny, Bobigny
  - SAMU Toulouse, Toulouse
- SAMU St-Denis de la Réunion, Saint-Denis, Reunion

REFERENCES:
- [Background] Jones JS, Johnson K, McNinch M. Age as a risk factor for inadequate emergency department analgesia. Am J Emerg Med. 1996 Mar;14(2):157-60. doi: 10.1016/S0735-6757(96)90123-0. PMID 8924137
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Doan BD. [Aging of population and medical workforce: a prospective view of health care provision in France in the year 2025]. Cah Sociol Demogr Med. 2004 Apr-Jun;44(2):243-66. French. PMID 15241964
- [Background] Strange GR, Chen EH. Use of emergency departments by elder patients: a five-year follow-up study. Acad Emerg Med. 1998 Dec;5(12):1157-62. doi: 10.1111/j.1553-2712.1998.tb02688.x. PMID 9864128